CLINICAL TRIAL: NCT00960518
Title: Combination Therapy With TACE and Adefovir Compared With TACE Alone for HBV-related Unresectable Hepatocellular Carcinoma
Brief Title: TACE and Adefovir Compared With Transarterial Chemoembolization (TACE) Alone for Hepatitis B Virus (HBV)-Related Unresectable Hepatocellular Carcinoma (HCC)
Acronym: TACE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Collaborators: Interventional Radiology Research Group, Shanghai Radiology Society (Unknown)
Responsible Party: Shanghai 10th Hospital, Tongji University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHDSYY20090725
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Hepatitis B Virus; Hepatocellular Carcinoma
Keywords: HBV-related unresectable HCC; TACE; adefovir; recurrence rate
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular | interventions — adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE (Placebo Comparator): An emulsion that consisted of 50 mg of cisplatin and 10 mL of lipiodol at a volume ratio of 1:1 was injected into the blood supply artery of the tumor under fluoroscopic guidance. The injection could be slowed or discontinued if retrograde flow occurred. Embolization was subsequently performed with granules of gelatin sponge particles.
  Interventions: Procedure: TACE
- TACE+adefovir (Experimental): patients received adefovir, at a dose of 10 mg daily after TACE treatment, for 48 weeks
  Interventions: Drug: adefovir

INTERVENTIONS:
Drug: adefovir — adefovir at 10 mg daily for 48 weeks
  Arms: TACE+adefovir
Procedure: TACE — An emulsion that consisted of 50 mg of cisplatin and 10 mL of lipiodol at a volume ratio of 1:1 was injected into the blood supply artery of the tumor under fluoroscopic guidance. The injection could be slowed or discontinued if retrograde flow occurred. Embolization was subsequently performed with granules of gelatin sponge particles.
  Arms: TACE

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most prevalent malignancies in China, and approximately 90% of the patients with HCC are also infected with hepatitis B virus (HBV). For patients with unresectable disease, the goal of palliative treatment is to control symptoms and prolong survival. Transarterial chemoembolization (TACE) using iodized oil and chemotherapeutic agents combines the effect of targeted chemotherapy with that of ischemic necrosis induced by arterial embolization. It can be administered repeatedly and can prolong survival in patients with unresectable hypervascular HCC. The long-term prognosis, however, remains guarded because of frequent development of locoregional tumor recurrence, which, together with concomitant hepatic decompensation, is the main cause of death. Adefovir works by blocking reverse transcriptase, an enzyme that is crucial for the hepatitis B virus (HBV) to reproduce in the body. Based on these results, the investigators conducted a randomized controlled trial to test the hypothesis that adefovir treatment would reduce or postpone the recurrence rate and improve the overall survival rate in patients after TACE treatment of HBV-related unresectable HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most prevalent malignancies in China, and approximately 90% of the patients with HCC are also infected with hepatitis B virus (HBV). Until now, no standard therapy has been established for treatment of hepatocellular carcinoma. For patients with unresectable disease, the goal of palliative treatment is to control symptoms and prolong survival. Transarterial chemoembolization (TACE) using iodized oil and chemotherapeutic agents combines the effect of targeted chemotherapy with that of ischemic necrosis induced by arterial embolization. It can be administered repeatedly and can prolong survival in patients with unresectable hypervascular HCC. The long-term prognosis, however, remains guarded because of frequent development of locoregional tumor recurrence, which, together with concomitant hepatic decompensation, is the main cause of death. Recurrence in the liver remnant may originate from metastasis from the primary tumor or multicentric new primaries in a cirrhotic liver.

Adefovir works by blocking reverse transcriptase, an enzyme that is crucial for the hepatitis B virus (HBV) to reproduce in the body. It is approved for the treatment of chronic hepatitis B in adults with evidence of active viral replication and either evidence of persistent elevations in serum aminotransferases (primarily ALT) or histologically active disease. The main benefit of adefovir over lamivudine (the first NRTI approved for the treatment of hepatitis B) is that it takes a much longer period of time before the virus develops resistance to it. Adefovir dipivoxil contains two pivaloyloxymethyl units, making it a prodrug form of Adefovir.

Based on these results, the investigators conducted a randomized controlled trial to test the hypothesis that adefovir treatment would reduce or postpone the recurrence rate and improve the overall survival rate in patients after TACE treatment of HBV-related unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* age:20-75 years old
* with a clinical diagnosis of primary liver cancer, with HBsAg positive,without any therapy for tumor
* single lesion with a diameter >6.5 cm,or multiple lesions locating within half liver or adjacent three lobe
* estimated liver remnant volume ≤40%
* with a liver function of Child-Pugh class A,and ALT≤80IU/l.

Exclusion Criteria:

* reject to attend
* portal vein trunk has been compressed by tumor
* diffuse type cancer or with extensive cancer thrombus in main branches of PV,HV,IVC or bile duct
* with extrahepatic metastasis
* with obvious portal hypertension (with moderate to severe varix in esophagus and/or gastric fundus, enlarged spleen,WBC<4×109／L, PLT<80×109／L)
* with diabetes
* allergy to iodine

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
the progression free survival (PFS) | 3 months

SECONDARY OUTCOMES:
the rate of overall survival | 1, 3, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Maoquan Li, MD, PhD, Study Chair — Interventional Radiology Research Group, Shanghai Radiology Society
Locations (2):
- China (2):
  - The Fourth Affiliated Hospital of Haerbin Medical University, Ha'er'bin, Heilongjiang
  - Shanghai 10th Hospital of Tongji University, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Li M, Lu C, Cheng J, Zhang J, Cao C, Xu J, Xu J, Pan H, Zhong B, Tucker S, Wang D. Combination therapy with transarterial chemoembolization and interferon-alpha compared with transarterial chemoembolization alone for hepatitis B virus related unresectable hepatocellular carcinoma. J Gastroenterol Hepatol. 2009 Aug;24(8):1437-44. doi: 10.1111/j.1440-1746.2009.05863.x. Epub 2009 May 28. PMID 19486255